CLINICAL TRIAL: NCT06888336
Title: Yoga Nidra Meditation for Insomnia and Posttraumatic Stress Symptoms: A Randomized-Controlled Feasibility Study
Brief Title: Yoga Nidra for Insomnia and Posttraumatic Stress Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 26303/002; ZIAMH002962 (NIH)
Record Dates: First submitted 2025-03-06; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Posttraumatic Stress Disorder (PTSD); Insomnia; Stressor, Psychological; Psychological Trauma
Keywords: randomized controlled trial; meditation; PTSD; insomnia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Sleep Initiation and Maintenance Disorders; Stress, Psychological; Psychological Trauma

STUDY DESIGN:
Intervention Model Description: Three-arm parallel assignment
Who Masked: Participant
Masking Description: Participants will be blinded to the presence of two different yoga nidra groups (high-dose and low-dose) during their participation in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yoga nidra (30 minutes each day) (Experimental): Participants will listen to ~30-minute yoga nidra meditation recordings every day for 8 weeks.
  Interventions: Behavioral: Yoga nidra (full)
- Yoga nidra (one 30-minute session/week, six 10-minute sessions/week) (Experimental): For 8 weeks, participants will be asked to listen to one ~30-minute yoga nidra meditation recording per week and six ~10-minute meditation recordings per week.
  Interventions: Behavioral: Yoga nidra (brief)
- Waitlist Control (No Intervention): During the intervention period, waitlist participants will not receive an intervention. At the end of Week 10, participants will be randomly assigned to low-dose yoga nidra or high-dose yoga nidra intervention for following the 8-week period.

INTERVENTIONS:
Behavioral: Yoga nidra (full) — The intervention consists of remotely delivered audio recordings (~30 minute length) of iRest yoga nidra meditation instructions that participants will be asked to listen to daily for 8 weeks, for a total listening time of about 3.5 hours each week. The yoga nidra practices will be in the tradition of iRest. They will include the following sections: intention setting, articulating a heartfelt desire, inner resource, body sensing, breath sensing, emotion and cognition sensing and opposites, welcoming joy, witnessing awareness, and integration. Each week includes an additional brief (~2-5 minute) introduction to one of the iRest yoga nidra sections. Participants will be asked to lie on a lightly cushioned surface when listening to the practices.
  Participants are informed that they may opt to listen to the recordings more often but are instructed to listen to the recordings at least once per day.
  Other Names: iRest
  Arms: Yoga nidra (30 minutes each day)
Behavioral: Yoga nidra (brief) — The intervention will consist of remotely delivered audio recordings of yoga nidra meditation instructions. Participants will be asked to listen to one ~30-minute practice and six ~10-minute practices per week (total listening time of ~1.5 hours each week) for 8 weeks. The yoga nidra practices will be in the tradition of iRest. They will include the following sections: intention setting, articulating a heartfelt desire, inner resource, body sensing, breath sensing, emotion and cognition sensing and opposites, welcoming joy, witnessing awareness, and integration. Each week includes an additional brief (2-5 minute) introduction to one of the iRest yoga nidra sections. Participants will be asked to lie on a lightly cushioned surface when listening to the practices.
  Participants are informed that they may opt to listen to the recordings more than once a day but are instructed to listen to the 30-minute recording once per week and the 10-minute meditations the other 6 days of the week.
  Other Names: iRest
  Arms: Yoga nidra (one 30-minute session/week, six 10-minute sessions/week)

SUMMARY:
This randomized feasibility study is designed to investigate the feasibility of recruitment and delivery of two variations (brief; full) of a virtual Integrative Restoration (iRest) yoga nidra meditation intervention in stressor- or trauma-exposed participants with insomnia and posttraumatic stress symptoms, compared to a waitlist control group. Feasibility will also be examined for data collection (daily sleep diaries and PTSD symptom surveys) and at-home polysomnography (PSG) study completion prior to and following the intervention. Feasibility measures will include study retention and-for the two yoga nidra groups-adherence to study protocol, and acceptability of the intervention will be assessed qualitatively, in semi-structured interviews, and quantitatively, with the Client Satisfaction Questionnaire, following the intervention. Acceptability of the daily surveys will also be assessed quantitatively.

Preliminary efficacy of the interventions on the primary treatment outcomes of insomnia and PTSD symptoms and symptom clusters will be assessed. Secondary outcomes include changes in specific sleep architecture assessed in an at-home polysomnogram (sleep stages, including stage N3 percentage, sleep spindles, rapid eye movement (REM) theta, total sleep time, wake after sleep onset time, sleep onset latency, sleep efficiency), daily sleep characteristics (total sleep time, sleep onset latency, wake after sleep onset time, sleep quality), daily PTSD symptoms, and mindfulness. Exploratory outcomes include sleep quality, experiential avoidance, emotion regulation, self-compassion, depression, anxiety, and nightmares.

DETAILED DESCRIPTION:
Participants will be randomly assigned to 1 of three groups: two remote yoga nidra interventions will be compared to a waitlist control group. The yoga nidra groups will be as follows: a high-dose condition in which participants will be instructed to engage in yoga nidra practice by listening to ~30-minute recordings every day for 8 weeks, and a low-dose condition in which participants will be instructed to engage in yoga nidra practice by listening to ~10-minute recordings 6 days per week and a ~30-minute recording one day per week for 8 weeks. The yoga nidra recordings are comprised of Integrative Restoration (iRest) yoga nidra scripts. Participants will be given the opportunity to listen to their provided recordings as often as they would like during the intervention. Frequency of practice sessions will be tracked on the website and recorded by participants in their daily surveys. In Week 10, participants in the waitlist control group will be randomly assigned to either low-dose or high-dose yoga nidra and given access to the recordings over the 8 weeks following the second PSG.

Daily PTSD symptoms and sleep will be recorded for two weeks prior to the intervention (baseline weeks) and throughout the intervention. At-home polysomnography will be completed immediately prior to the intervention (Week 2) and immediately following the intervention (Week 10), and questionnaires will be completed during the in-lab electrode application and removal sessions for the at-home polysomnography. During the in-lab sessions, resting state electroencephalography (EEG), heart rate variability (HRV), and skin conductance levels will also be recorded. Follow-up questionnaires will be administered to all participants 8 weeks after the second sleep study (Week 18) to assess primary treatment outcomes and mindfulness in waitlist participants after the intervention and maintenance of primary treatment outcomes and mindfulness following the intervention in yoga nidra high- and low-dose participants.

ELIGIBILITY:
Inclusion Criteria:

* Endorses experiencing at least one lifetime very stressful or traumatic event that still distresses them
* Score of 13 or higher on the 8-item PCL-5
* Scoring 15 or higher on the Insomnia Severity Index, indicating the presence of moderate to severe insomnia
* Being able and willing to listen to online yoga nidra audio recordings that may each be up to 35 minutes long daily for 8 weeks
* Being willing to monitor sleep and PTSD symptoms for 10 weeks
* Normal or corrected to normal hearing and vision
* Fluent in English
* Reliable daily access to the internet Between the ages of 18 and 35
* Between the ages of 18 and 35
* Reliable daily access to the internet
* Willing to refrain from ingesting caffeine, alcohol, and recreational drugs the day of the sleep studies
* Currently receiving or seeking treatment for alcoholism or a substance abuse disorder

Exclusion Criteria:

* History of schizophrenia, psychotic disorder, or bipolar disorder
* Current endorsement of suicidality (score of 2 or higher on Item 9 of the BDI-II)
* Currently receiving psychological treatment for any mental health disorder
* Current diagnosis of any sleep disorder, excluding insomnia or nightmare disorder
* Currently taking benzodiazepines, nonbenzodiazepine receptor agonists, orexin agonists or antagonists, antiseizure medication, any medications for sleep
* Score of 5 or higher on STOP-BANG Questionnaire (indicating likelihood of moderate to severe obstructive sleep apnea)
* Previous adverse experience with meditation
* Current regular meditative practice (meditating once or more per month)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility: Participant Retention | From baseline to follow-up (Weeks 1-10, Week 10, Week 18)
  Retention will be quantified as percentage of participants that complete different levels of the acute protocol (i.e. ≤25%, 26-50%, 51-75%, > 75% of daily questionnaires, and second at-home PSG) and percentage that complete the follow-up questionnaires.
Feasibility: Adherence to Yoga Nidra Protocol | Throughout treatment (Week 2 to 10)
  Adherence will be quantified as percentage of participants that complete 1-7 sessions in each week. Also, a measure of 'quality of meditation' (assessed using the PQ-M for each reported meditation) will serve as an additional measure of adherence.

SECONDARY OUTCOMES:
Sleep Characteristics, Assessed in the At-home PSG | Change from baseline to post-treatment (Week 2; Week 10)
  At-home polysomnography will be used to measure sleep architecture. Sleep characteristics of interest include N3 percentage, Sleep onset latency, Wake after sleep onset time, Total sleep time, Sleep spindles, and REM theta.
Daily Sleep Characteristics | From baseline to end of treatment/waitlist period (Weeks 1 to 10)
  This will be assessed using the Consensus Sleep Diary - E, with an additional question administered in the morning to record number of nightmares experienced. Daily sleep characteristics will include: total sleep time, sleep onset latency, wake after sleep onset time, and number of nightmares.
Daily PTSD Symptom Severity | From baseline to end of treatment/waitlist period (Weeks 1 to 10)
  A daily version of the PCL-5 8-item version will be administered each day, for participants to complete shortly before going to bed. The PCL-5 8-item version is an abbreviated version of the full-length PCL-5, with 2 symptoms assessed for each symptom cluster and ratings on a 5-point Likert scale (0 = Not at all bothered, 4 = Very bothered).
PTSD Symptoms (PCL-5) | Change from baseline to end of treatment and follow-up (Week 2; 10; 18)
  The PTSD Checklist for the DSM-5 (PCL-5) is a self-report questionnaire used to assess severity of DSM-5 PTSD symptoms over the past month. It includes 20 items (5 per symptom cluster), each rated on a 5-point Likert scale (0 = Not at all bothered by, 4 = Extremely bothered by).
Insomnia Symptoms (ISI) | Change from baseline to end of treatment and follow-up (Week 2; Week 10; Week 18)
  The Insomnia Severity Index (ISI) is a 7-item questionnaires that assesses the severity of daytime and nighttime components of insomnia over the past two weeks. A 5-point Likert scale (0 = No problem, 4 = Very severe problem) is provided for each item, and scores range from 0 to 28, with higher scores indicating greater insomnia severity.
Mindfulness (FFMQ-15) | Change from baseline to end of treatment and follow-up (Week 2; Week 10; Week 18)
  The Five Facet Mindfulness Questionnaire, 15-item version (FFMQ-15) assesses five facets of mindfulness (Observing, Describing, Acting with Awareness, Nonjudging of Inner Experience, Nonreactivity to Inner Experience). Each item is rated from 1 to 5 ( 1 = Never or very rarely true; 5 = Very often or always true) according to what is generally true for the respondent, and there are 7 reverse-scored items. For all FFMQ-15 subscales, scores range from 3 to 15, with higher scores indicating greater mindfulness.
Acceptability of Intervention (CSQ) | Post-treatment (Week 10)
  The Client Satisfaction Questionnaire-8 (CSQ-8) is an 8-item measure of satisfaction with a treatment. Each item is rated on a 4-point Likert scale, in which "1" indicates the lowest level of satisfaction and "4" indicates the highest level of satisfaction.
Acceptability Ratings of Daily Surveys | Post-treatment/waitlist (Week 10)
  At conclusion of the daily monitoring period (Post-treatment/waitlist or Dropout), participants will respond to 10 questions intended to assess daily survey acceptability on a 7-point Likert scale (1 = Strongly Disagree; 7 = Strongly Agree) (adapted from Mintz et al., 2024).

OTHER OUTCOMES:
Experiential Avoidance (BEAQ) | Change from baseline to post-treatment (Week 2; Week 10)
  The Brief Experiential Avoidance Questionnaire (BEAQ) is a 15-item scale, abbreviated from the Multidimensional Experiential Avoidance Questionnaire (MEAQ). There are six subscales (Behavioral Avoidance, Distress Aversion, Procrastination, Distraction/Suppression, Repression/Denial, and Distress Endurance). Each item is rated on a 6-point Likert scale (1 = Strongly disagree; 6 = Strongly agree).
Nightmare Disorder Symptom Severity (NDI) | Change from baseline to post-treatment (Week 2; Week 10)
  The Nightmare Disorder Index (NDI) is a 5-item measure used to assess frequency, characteristics, distress, and impairment due to nightmares over the past month, according to DSM-5 criteria for nightmare disorder. Each item is assessed on a 5-point Likert scale from 0 to 4.
Sleep Quality (PSQI) | Change from baseline to post-treatment (Week 2; Week 10)
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item questionnaire used to assess sleep quality over the past month, with higher scores indicating worse sleep quality. A score of > 5 is typically considered to indicate poor sleep.
Emotion Regulation (ERQ-9) | Change from baseline to post-treatment (Week 2; Week 10)
  The Emotion Regulation Questionnaire-9 (ERQ-9) is a 9-item questionnaire used to assess tendency to use two emotion regulation strategies (reappraisal and suppression). Items are rated on a 7-point Likert scale from 1 (Strongly disagree) to 7 (Strongly agree).
Self-Compassion (SOCS-S) | Change from baseline to post-treatment (Week 2; Week 10)
  The Sussex-Oxford Compassion for the Self Scale (SOCS-S) is a 20-item questionnaire used to assess self-compassion. Each item is rated on a 5-point Likert scale (1 = Not at all true, 5 = Always true).
Depressive Symptoms (BDI-II) | Change from baseline to post-treatment (Week 2; Week 10)
  The Beck Depression Inventory-II (BDI-II) is a 21-item self-report questionnaire used to assess major depression symptoms over the past 2 weeks. Each item is rated on a Likert scale from 0 to 4, with higher scores indicating greater severity.
Anxiety Symptoms (STAI) | Change from baseline to post-treatment (Week 2; Week 10)
  The State Trait Anxiety Index, Form Y-2 (STAI) is a 20-item self-report questionnaire used to assess anxiety severity. Participants are asked to rate each item on a Likert scale from 1 to 4 (1 = Not at all, 4 = Very much so) to indicate how they generally feel.
Qualitative Feedback | Post-treatment (Week 10)
  Qualitative feedback on the acceptability, content, and structure of the intervention will be obtained during semi-structured interviews, which will be conducted with yoga nidra (high dose and low dose) participants in person after the treatment period.
Daily Intrusive Memories | From baseline to end of treatment/waitlist period (Weeks 1 to 10)
  The number of intrusive memories and (if any) their distress and vividness, as rated on a 7-point Likert scale (1 = Not at all; 7 = Extremely), will be recorded by participants each day before going to bed.
Mindfulness Practice Quality (PQ-M) | Throughout treatment (Weeks 2 to 10)
  For participants in the yoga nidra groups, Practice Quality-Mindfulness (PQ-M; Del Re et al., 2022), a 6-item questionnaire, will be used to monitor meditation practice quality daily throughout the intervention. For each statement, participants are asked to indicate the approximate percentage of time that their meditation experience reflected the statement. The PQ-M is comprised of two components: receptivity and attention.
Heart Rate Variability (HRV) | Change from baseline to post-treatment (Week 2; Week 10)
  Heart rate variability will be derived from resting-state heart rate, as measured before and after the intervention period.
Skin Conductance Level (SCL) | Change from baseline to post-treatment (Week 2; Week 10)
  Resting-state skin conductance will be measured with the Empatica EmbracePlus wristbands before and after the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Sunjeev Kamboj, PhD, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified demographic, questionnaire, and physiological participant data will be shared.
Supporting Information: Study Protocol
Time Frame: Anticipated to begin within 18 months of completion of data collection
Access Criteria: Data will be made available through controlled access with the National Sleep Research Repository (NSRR), which aims to make data available indefinitely.